CLINICAL TRIAL: NCT03368053
Title: Long-term Immunogenicity of the HIV gp120-NefTat/AS01B Vaccine (GSK SB732461)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201606
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2019-11-18 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: gp120; HIV infections; RV144; gp120-NefTat/AS01B vaccine candidate; V1V2
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Descriptive mono-centric study with one single group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GSKSB732461 Group (Experimental): Healthy HIV uninfected volunteers who participated in study PRO HIV-002 between February 2003 and February 2005 and who were vaccinated with at least 3 doses of the GSKSB732461 vaccine candidate in the PRO-HIV-002 study.
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood samples will be taken during the single study visit at Year 14 for the assessment of: HIV testing, antibody determination, cell mediated immune (CMI) responses and exploratory characterisation.

SUMMARY:
The purpose of this study is to evaluate the long-term persistence of binding antibody responses against V1V2 and gp120 in subjects who were vaccinated with the envelope glycoprotein 120 (gp120)-negative factor (Nef)Tat/ Adjuvant System 01B (AS01B) (GSKSB732461) vaccine candidate. Other immune parameters like the HIV-specific cluster of differentiation (CD4+) T cell and CD8+ T cell responses will also be evaluated.

DETAILED DESCRIPTION:
GlaxoSmithKline (GSK) contributes to the public-private pox-protein partnership (P5) which is currently assessing the safety, immunogenicity and clinical efficacy of a prime-boost regimen aimed at preventing HIV transmission (http://www.hvtn.org/en.html). The booster component of the candidate vaccine used in this program consists of two gp120 clade C proteins administered with an adjuvant. In order to inform the selection of the adjuvant in future studies, data on long-term persistence of immunity after vaccination with gp120/AS01 would prove useful. The present study was designed to address this question using a cohort of volunteers vaccinated several years ago with a candidate vaccine containing gp120 and AS01.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* A subject who has received at least 3 doses of the gp120-NefTat/AS01B (GSKSB732461) vaccine candidate in GSK Biologicals-sponsored PRO HIV-002 study.

Exclusion Criteria:

* Use of any investigational or non-registered product during 30 days prior to study enrolment.
* History of HIV-1 or HIV-2 infection.
* Participation to another clinical trial of an investigational HIV vaccine between study PRO HIV-002 and the present study.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting one month preceding this study. For corticosteroids, this will mean prednisone higher than or equal to (≥) 20 mg/day . Inhaled and topical steroids are allowed.
* Administration of cytotoxic medication within 6 months preceding this study.
* History of daily, long-term immunosuppressive medication between study PRO HIV-002 and the present study.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before enrolment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition other than HIV disease, based on medical history and physical examination between study PRO HIV-002 and the present study.
* Past administration of an investigational vaccine containing AS01 other than the gp120-NefTat/AS01B (GSKSB732461) vaccine administered in PRO HIV-002 study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20331

REFERENCES:
- [Background] Van Der Meeren O, Jongert E, Seaton KE, Koutsoukos M, Aerssens A, Brackett C, Debois M, Janssens M, Leroux-Roels G, Mesia Vela D, Sawant S, Yates NL, Tomaras GD, Leroux-Roels I, Roman F. Persistence of vaccine-elicited immune response up to 14 years post-HIV gp120-NefTat/AS01B vaccination. Vaccine. 2020 Feb 11;38(7):1678-1689. doi: 10.1016/j.vaccine.2019.12.058. Epub 2020 Jan 10. PMID 31932137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one Centre in Belgium.
Pre-assignment Details: A total of 36 subjects were enrolled in the study. Those subjects received at least three doses of the GSKSB732461 vaccine candidate in GSK-sponsored 732461/002 (PRO HIV-002) study.
Period: Overall Study
Arm/Group | GSKSB732461 Group
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE - CAUCASIAN / EUROPEAN HERITAGE | 35
  BLACK OR AFRICAN AMERICAN | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-V1V2 Total Immunoglobulin G (IgG) Binding Antibody Multiplex Assay (BAMA) Response Call
Description: To comply with BAMA methodology and terminology, the wording "BAMA response call status" was used instead of "seropositivity" in the analysis. Compared to baseline result (Day 0), a sample is called "positive" for a given analyte if the response magnitude is equal to or above (≥) the analyte specific cutoff from all baseline samples in the study (where the cutoff is the 95th percentile of the baseline response, or 100, whichever is higher) OR ≥3 times the response magnitude as compared to the sample specific baseline. The C.1086C_V1_V2 Tags strain was not part of any breadth panel. Due to low or infrequent response, or undetectable levels of response among the breadth panel strains, some additional strains, not part of the breadth panels, were also analyzed.
Time Frame: At Day 182, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: Analysis was performed on the Per-Protocol cohort for immunogenicity which included all subjects from the Total cohort who met all eligibility criteria, and who presented a negative HIV-RNA test at Y14.
Measure: Count of Participants; unit: Participants
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 27
Participants
  gp70-001428.2.42 strain, at Day 182: number analyzed (Participants) | 26
  gp70-001428.2.42 strain, at Day 182 | 25
  gp70-001428.2.42 strain, at Day 672 | 15
  gp70-001428.2.42 strain, at Year 14: number analyzed (Participants) | 23
  gp70-001428.2.42 strain, at Year 14 | 8
  gp70-191084_B7 strain, at Day 182: number analyzed (Participants) | 26
  gp70-191084_B7 strain, at Day 182 | 20
  gp70-191084_B7 strain, at Day 672 | 12
  gp70-191084_B7 strain, at Year 14: number analyzed (Participants) | 23
  gp70-191084_B7 strain, at Year 14 | 9
  gp70-62357.14 strain, at Day 182: number analyzed (Participants) | 26
  gp70-62357.14 strain, at Day 182 | 12
  gp70-62357.14 strain, at Day 672 | 1
  gp70-62357.14 strain, at Year 14: number analyzed (Participants) | 23
  gp70-62357.14 strain, at Year 14 | 0
  gp70-700010058 strain, at Day 182: number analyzed (Participants) | 26
  gp70-700010058 strain, at Day 182 | 26
  gp70-700010058 strain, at Day 672: number analyzed (Participants) | 26
  gp70-700010058 strain, at Day 672 | 19
  gp70-700010058 strain, at Year 14: number analyzed (Participants) | 23
  gp70-700010058 strain, at Year 14 | 13
  gp70-7060101641 strain, at Day 182: number analyzed (Participants) | 26
  gp70-7060101641 strain, at Day 182 | 18
  gp70-7060101641 strain, at Day 672 | 9
  gp70-7060101641 strain, at Year 14: number analyzed (Participants) | 23
  gp70-7060101641 strain, at Year 14 | 4
  gp70-96ZM651.02 strain, at Day 182: number analyzed (Participants) | 26
  gp70-96ZM651.02 strain, at Day 182 | 21
  gp70-96ZM651.02 strain, at Day 672: number analyzed (Participants) | 26
  gp70-96ZM651.02 strain, at Day 672 | 4
  gp70-96ZM651.02 strain, at Year 14: number analyzed (Participants) | 23
  gp70-96ZM651.02 strain, at Year 14 | 2
  gp70-BF1266_431a strain, at Day 182: number analyzed (Participants) | 26
  gp70-BF1266_431a strain, at Day 182 | 24
  gp70-BF1266_431a strain, at Day 672: number analyzed (Participants) | 26
  gp70-BF1266_431a strain, at Day 672 | 16
  gp70-BF1266_431a strain, at Year 14: number analyzed (Participants) | 23
  gp70-BF1266_431a strain, at Year 14 | 11
  gp70-BJOX002000.03.2 strain, at Day 182: number analyzed (Participants) | 26
  gp70-BJOX002000.03.2 strain, at Day 182 | 24
  gp70-BJOX002000.03.2 strain, at Day 672 | 14
  gp70-BJOX002000.03.2 strain, at Year 14: number analyzed (Participants) | 22
  gp70-BJOX002000.03.2 strain, at Year 14 | 6
  gp70-C2101.c01 strain, at Day 182: number analyzed (Participants) | 26
  gp70-C2101.c01 strain, at Day 182 | 20
  gp70-C2101.c01 strain, at Day 672: number analyzed (Participants) | 26
  gp70-C2101.c01 strain, at Day 672 | 12
  gp70-C2101.c01 strain, at Year 14: number analyzed (Participants) | 22
  gp70-C2101.c01 strain, at Year 14 | 8
  gp70-CAP210.2.00.E8 strain, at Day 182: number analyzed (Participants) | 26
  gp70-CAP210.2.00.E8 strain, at Day 182 | 26
  gp70-CAP210.2.00.E8 strain, at Day 672 | 15
  gp70-CAP210.2.00.E8 strain, at Year 14: number analyzed (Participants) | 23
  gp70-CAP210.2.00.E8 strain, at Year 14 | 7
  gp70-CM244.ec1 strain, Day 182: number analyzed (Participants) | 26
  gp70-CM244.ec1 strain, Day 182 | 22
  gp70-CM244.ec1 strain, at Day 672: number analyzed (Participants) | 26
  gp70-CM244.ec1 strain, at Day 672 | 13
  gp70-CM244.ec1 strain, at Year 14: number analyzed (Participants) | 23
  gp70-CM244.ec1 strain, at Year 14 | 7
  gp70-Ce1086_B2 strain, at Day 182: number analyzed (Participants) | 26
  gp70-Ce1086_B2 strain, at Day 182 | 23
  gp70-Ce1086_B2 strain, at Day 672 | 14
  gp70-Ce1086_B2 strain, at Year 14: number analyzed (Participants) | 23
  gp70-Ce1086_B2 strain, at Year 14 | 6
  gp70-RHPA4259.7 strain, at Day 182: number analyzed (Participants) | 26
  gp70-RHPA4259.7 strain, at Day 182 | 22
  gp70-RHPA4259.7 strain, at Day 672: number analyzed (Participants) | 26
  gp70-RHPA4259.7 strain, at Day 672 | 9
  gp70-RHPA4259.7 strain, at Year 14: number analyzed (Participants) | 23
  gp70-RHPA4259.7 strain, at Year 14 | 2
  gp70-TT31P.2F10.2792 strain, at Day 182: number analyzed (Participants) | 26
  gp70-TT31P.2F10.2792 strain, at Day 182 | 26
  gp70-TT31P.2F10.2792 strain, at Day 672: number analyzed (Participants) | 26
  gp70-TT31P.2F10.2792 strain, at Day 672 | 18
  gp70-TT31P.2F10.2792 strain, at Year 14: number analyzed (Participants) | 23
  gp70-TT31P.2F10.2792 strain, at Year 14 | 10
  gp70-TV1.21 strain, at Day 182: number analyzed (Participants) | 26
  gp70-TV1.21 strain, at Day 182 | 26
  gp70-TV1.21 strain, at Day 672 | 18
  gp70-TV1.21 strain, at Year 14: number analyzed (Participants) | 23
  gp70-TV1.21 strain, at Year 14 | 9
  gp70_B.CaseA strain, at Day 182: number analyzed (Participants) | 26
  gp70_B.CaseA strain, at Day 182 | 26
  gp70_B.CaseA strain, at Day 672: number analyzed (Participants) | 26
  gp70_B.CaseA strain, at Day 672 | 21
  gp70_B.CaseA strain, at Year 14: number analyzed (Participants) | 23
  gp70_B.CaseA strain, at Year 14 | 12
  C.1086C_V1_V2 Tags strain, at Day 182 | 19
  C.1086C_V1_V2 Tags strain, at Day 672 | 5
  C.1086C_V1_V2 Tags strain, at Year 14: number analyzed (Participants) | 23
  C.1086C_V1_V2 Tags strain, at Year 14 | 3

2. Primary Outcome: Anti-V1V2 Total IgG Antibody BAMA Response Magnitude
Description: Whenever results were provided as "Mean Fluorescence Intensity (MFI)", the statistical outputs "BAMA response magnitude (MFI)" terminology is used instead of "concentrations/titres". The C.1086C_V1_V2 Tags strain was not part of any breadth panel. Due to low or infrequent response, or undetectable levels of response among the breadth panel strains, some additional strains, not part of the breadth panels, were also analyzed.
Time Frame: At Day 0, Day 182, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: MFI
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 32
MFI
  gp70-001428.2.42 strain, at Day 0: number analyzed (Participants) | 28
  gp70-001428.2.42 strain, at Day 0 | 1.3 [0.9 to 1.9]
  gp70-001428.2.42 strain, at Day 182: number analyzed (Participants) | 30
  gp70-001428.2.42 strain, at Day 182 | 5444.9 [2974.9 to 9965.9]
  gp70-001428.2.42 strain, at Day 672: number analyzed (Participants) | 31
  gp70-001428.2.42 strain, at Day 672 | 147.5 [41.1 to 529.7]
  gp70-001428.2.42 strain, at Year 14: number analyzed (Participants) | 28
  gp70-001428.2.42 strain, at Year 14 | 29.5 [9.4 to 92.9]
  gp70-191084_B7 strain, at Day 0: number analyzed (Participants) | 28
  gp70-191084_B7 strain, at Day 0 | 1.4 [0.9 to 2.1]
  gp70-191084_B7 strain, at Day 182: number analyzed (Participants) | 30
  gp70-191084_B7 strain, at Day 182 | 1272.5 [308.2 to 5254.8]
  gp70-191084_B7 strain, at Day 672: number analyzed (Participants) | 31
  gp70-191084_B7 strain, at Day 672 | 98.2 [22.6 to 426.5]
  gp70-191084_B7 strain, at Year 14: number analyzed (Participants) | 28
  gp70-191084_B7 strain, at Year 14 | 28.4 [6.6 to 122.9]
  gp70-62357.14 strain, at Day 0: number analyzed (Participants) | 28
  gp70-62357.14 strain, at Day 0 | 1.4 [0.8 to 2.4]
  gp70-62357.14 strain, at Day 182: number analyzed (Participants) | 30
  gp70-62357.14 strain, at Day 182 | 33.4 [11.3 to 98.5]
  gp70-62357.14 strain, at Day 672: number analyzed (Participants) | 31
  gp70-62357.14 strain, at Day 672 | 2.0 [1.0 to 3.8]
  gp70-62357.14 strain, at Year 14: number analyzed (Participants) | 28
  gp70-62357.14 strain, at Year 14 | 1.2 [0.9 to 1.7]
  gp70-700010058 strain, at Day 0: number analyzed (Participants) | 28
  gp70-700010058 strain, at Day 0 | 1.4 [0.9 to 2.1]
  gp70-700010058 strain, at Day 182: number analyzed (Participants) | 30
  gp70-700010058 strain, at Day 182 | 18048.6 [12831.6 to 25386.6]
  gp70-700010058 strain, at Day 672: number analyzed (Participants) | 30
  gp70-700010058 strain, at Day 672 | 925.0 [264.5 to 3235.1]
  gp70-700010058 strain, at Year 14: number analyzed (Participants) | 28
  gp70-700010058 strain, at Year 14 | 130.1 [36.7 to 461.3]
  gp70-7060101641 strain, at Day 0: number analyzed (Participants) | 28
  gp70-7060101641 strain, at Day 0 | 1.2 [0.9 to 1.7]
  gp70-7060101641 strain, at Day 182: number analyzed (Participants) | 30
  gp70-7060101641 strain, at Day 182 | 353.7 [108.0 to 1157.8]
  gp70-7060101641 strain, at Day 672: number analyzed (Participants) | 31
  gp70-7060101641 strain, at Day 672 | 23.5 [6.8 to 81.0]
  gp70-7060101641 strain, at Year 14: number analyzed (Participants) | 28
  gp70-7060101641 strain, at Year 14 | 13.4 [4.4 to 40.5]
  gp70-96ZM651.02 strain, at Day 0: number analyzed (Participants) | 28
  gp70-96ZM651.02 strain, at Day 0 | 1.7 [1.0 to 3.0]
  gp70-96ZM651.02 strain, at Day 182: number analyzed (Participants) | 30
  gp70-96ZM651.02 strain, at Day 182 | 777.3 [286.8 to 2106.5]
  gp70-96ZM651.02 strain, at Day 672: number analyzed (Participants) | 30
  gp70-96ZM651.02 strain, at Day 672 | 11.2 [3.7 to 33.5]
  gp70-96ZM651.02 strain, at Year 14: number analyzed (Participants) | 28
  gp70-96ZM651.02 strain, at Year 14 | 4.5 [1.9 to 10.6]
  gp70-BF1266_431a strain, at Day 0: number analyzed (Participants) | 28
  gp70-BF1266_431a strain, at Day 0 | 1.3 [0.9 to 2.1]
  gp70-BF1266_431a strain, at Day 182: number analyzed (Participants) | 30
  gp70-BF1266_431a strain, at Day 182 | 7838.7 [3122.7 to 19676.7]
  gp70-BF1266_431a strain, at Day 672: number analyzed (Participants) | 30
  gp70-BF1266_431a strain, at Day 672 | 414.6 [90.9 to 1890.9]
  gp70-BF1266_431a strain, at Year 14: number analyzed (Participants) | 28
  gp70-BF1266_431a strain, at Year 14 | 94.7 [22.0 to 408.3]
  gp70-BJOX002000.03.2 strain, at Day 0: number analyzed (Participants) | 28
  gp70-BJOX002000.03.2 strain, at Day 0 | 1.3 [0.9 to 1.8]
  gp70-BJOX002000.03.2 strain, at Day 182: number analyzed (Participants) | 30
  gp70-BJOX002000.03.2 strain, at Day 182 | 4033.1 [1722.3 to 9444.1]
  gp70-BJOX002000.03.2 strain, at Day 672: number analyzed (Participants) | 31
  gp70-BJOX002000.03.2 strain, at Day 672 | 113.7 [30.5 to 424.5]
  gp70-BJOX002000.03.2 strain, at Year 14: number analyzed (Participants) | 27
  gp70-BJOX002000.03.2 strain, at Year 14 | 22.3 [6.6 to 75.3]
  gp70-C2101.c01 strain, at Day 0: number analyzed (Participants) | 28
  gp70-C2101.c01 strain, at Day 0 | 1.3 [0.9 to 1.6]
  gp70-C2101.c01 strain, at Day 182: number analyzed (Participants) | 30
  gp70-C2101.c01 strain, at Day 182 | 1454.2 [356.9 to 5925.2]
  gp70-C2101.c01 strain, at Day 672: number analyzed (Participants) | 30
  gp70-C2101.c01 strain, at Day 672 | 85.0 [17.1 to 422.6]
  gp70-C2101.c01 strain, at Year 14: number analyzed (Participants) | 27
  gp70-C2101.c01 strain, at Year 14 | 28.7 [6.2 to 131.8]
  gp70-CAP210.2.00.E8 strain, at Day 0: number analyzed (Participants) | 28
  gp70-CAP210.2.00.E8 strain, at Day 0 | 1.2 [0.9 to 1.6]
  gp70-CAP210.2.00.E8 strain, at Day 182: number analyzed (Participants) | 30
  gp70-CAP210.2.00.E8 strain, at Day 182 | 5862.5 [3157.3 to 10885.8]
  gp70-CAP210.2.00.E8 strain, at Day 672: number analyzed (Participants) | 31
  gp70-CAP210.2.00.E8 strain, at Day 672 | 150.2 [40.6 to 556.2]
  gp70-CAP210.2.00.E8 strain, at Year 14: number analyzed (Participants) | 28
  gp70-CAP210.2.00.E8 strain, at Year 14 | 32.9 [9.7 to 111.0]
  gp70-CM244.ec1 strain, at Day 0: number analyzed (Participants) | 28
  gp70-CM244.ec1 strain, at Day 0 | 1.6 [0.9 to 2.6]
  gp70-CM244.ec1 strain, at Day 182: number analyzed (Participants) | 30
  gp70-CM244.ec1 strain, at Day 182 | 2770.8 [1057.6 to 7259.5]
  gp70-CM244.ec1 strain, at Day 672: number analyzed (Participants) | 30
  gp70-CM244.ec1 strain, at Day 672 | 98.6 [22.7 to 429.2]
  gp70-CM244.ec strain, at Year 14: number analyzed (Participants) | 28
  gp70-CM244.ec strain, at Year 14 | 33.0 [8.7 to 124.8]
  gp70-Ce1086_B2 strain, at Day 0: number analyzed (Participants) | 28
  gp70-Ce1086_B2 strain, at Day 0 | 1.3 [0.9 to 2.0]
  gp70-Ce1086_B2 strain, at Day 182: number analyzed (Participants) | 30
  gp70-Ce1086_B2 strain, at Day 182 | 2336.9 [889.9 to 6136.8]
  gp70-Ce1086_B2 strain, at Day 672: number analyzed (Participants) | 31
  gp70-Ce1086_B2 strain, at Day 672 | 82.8 [20.9 to 328.6]
  gp70-Ce1086_B2 strain, at Year 14: number analyzed (Participants) | 28
  gp70-Ce1086_B2 strain, at Year 14 | 23.4 [6.6 to 83.3]
  gp70-RHPA4259.7 strain, at Day 0: number analyzed (Participants) | 28
  gp70-RHPA4259.7 strain, at Day 0 | 1.5 [0.9 to 2.4]
  gp70-RHPA4259.7 strain, at Day 182: number analyzed (Participants) | 30
  gp70-RHPA4259.7 strain, at Day 182 | 2033.8 [638.2 to 6481.8]
  gp70-RHPA4259.7 strain, at Day 672: number analyzed (Participants) | 30
  gp70-RHPA4259.7 strain, at Day 672 | 30.4 [8.9 to 103.9]
  gp70-RHPA4259.7 strain, at Year 14: number analyzed (Participants) | 28
  gp70-RHPA4259.7 strain, at Year 14 | 6.5 [2.5 to 17.1]
  gp70-TT31P.2F10.2792 strain, at Day 0: number analyzed (Participants) | 28
  gp70-TT31P.2F10.2792 strain, at Day 0 | 1.5 [0.9 to 2.4]
  gp70-TT31P.2F10.2792 strain, at Day 182: number analyzed (Participants) | 30
  gp70-TT31P.2F10.2792 strain, at Day 182 | 10998.7 [6967.0 to 17363.3]
  gp70-TT31P.2F10.2792 strain, at Day 672: number analyzed (Participants) | 30
  gp70-TT31P.2F10.2792 strain, at Day 672 | 312.7 [82.8 to 1181.0]
  gp70-TT31P.2F10.2792 strain, at Year 14: number analyzed (Participants) | 28
  gp70-TT31P.2F10.2792 strain, at Year 14 | 71.9 [20.9 to 247.8]
  gp70-TV1.21 strain, at Day 0: number analyzed (Participants) | 28
  gp70-TV1.21 strain, at Day 0 | 1.4 [0.9 to 2.2]
  gp70-TV1.21 strain, at Day 182: number analyzed (Participants) | 30
  gp70-TV1.21 strain, at Day 182 | 10684.4 [6527.9 to 17487.7]
  gp70-TV1.21 strain, at Day 672: number analyzed (Participants) | 31
  gp70-TV1.21 strain, at Day 672 | 382.4 [108.3 to 1350.5]
  gp70-TV1.21 strain, at Year 14: number analyzed (Participants) | 28
  gp70-TV1.21 strain, at Year 14 | 75.7 [21.6 to 265.4]
  gp70_B.CaseA strain, at Day 0: number analyzed (Participants) | 28
  gp70_B.CaseA strain, at Day 0 | 1.7 [0.9 to 3.1]
  gp70_B.CaseA strain, at Day 182: number analyzed (Participants) | 30
  gp70_B.CaseA strain, at Day 182 | 21647.6 [16859.7 to 27795.3]
  gp70_B.CaseA strain, at Day 672: number analyzed (Participants) | 30
  gp70_B.CaseA strain, at Day 672 | 1104.4 [327.0 to 3730.2]
  gp70_B.CaseA strain, at Year 14: number analyzed (Participants) | 28
  gp70_B.CaseA strain, at Year 14 | 166.6 [46.9 to 591.5]
  C.1086C_V1_V2 Tags strain, at Day 0: number analyzed (Participants) | 27
  C.1086C_V1_V2 Tags strain, at Day 0 | 1.2 [0.8 to 1.9]
  C.1086C_V1_V2 Tags strain, at Day 182 | 216.4 [76.9 to 609.1]
  C.1086C_V1_V2 Tags strain, at Day 672: number analyzed (Participants) | 31
  C.1086C_V1_V2 Tags strain, at Day 672 | 15.1 [5.8 to 39.6]
  C.1086C_V1_V2 Tags strain, at Year 14: number analyzed (Participants) | 27
  C.1086C_V1_V2 Tags strain, at Year 14 | 4.7 [2.0 to 11.5]

3. Primary Outcome: Number of Subjects With Anti-V1V2 Subtypes Range: IgG1, IgG2, IgG3 and IgG4 Response Call
Description: To comply with BAMA methodology and terminology, the wording "BAMA response call status" was used instead of "seropositivity" in the analysis. Compared to baseline result (Day 0), a sample is called "positive" for a given analyte if the response magnitude is equal to or above (≥) the analyte specific cutoff from all baseline samples in the study (where the cutoff is the 95th percentile of the baseline response, or 100, whichever is higher) OR ≥3 times the response magnitude as compared to the sample specific baseline. Antigen IgG3 was assessed for all strains. Antigens IgG1, IgG2 and IgG4 were assessed only for C.1086C_V1_V2 Tags strain that was not part of any breadth panel. Due to low or infrequent response, or undetectable levels of response among the breadth panel strains, some additional strains, not part of the breadth panels, were also analyzed.
Time Frame: At Day 182, Day 672 historical time point of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 29
Participants
  gp70-001428.2.42 IgG3 strain, at Day 182 | 2
  gp70-001428.2.42 IgG3 strain, at Day 672 | 0
  gp70-001428.2.42 IgG3 strain, at Year 14 | 0
  gp70-191084_B7 IgG3 strain, at Day 182 | 2
  gp70-191084_B7 IgG3 strain, at Day 672 | 1
  gp70-191084_B7 IgG3 strain, at Year 14 | 0
  gp70-62357.14 IgG3 strain, at Day 182 | 0
  gp70-62357.14 IgG3 strain, at Day 672 | 0
  gp70-62357.14 IgG3 strain, at Year 14 | 0
  gp70-700010058 IgG3 strain, at Day 182 | 3
  gp70-700010058 IgG3 strain, at Day 672 | 0
  gp70-700010058 IgG3 strain, at Year 14 | 0
  gp70-7060101641 IgG3 strain, at Day 182 | 0
  gp70-7060101641 IgG3 strain, at Day 672 | 0
  gp70-7060101641 IgG3 strain, at Year 14 | 0
  gp70-96ZM651.02 IgG3 strain, at Day 182 | 0
  gp70-96ZM651.02 IgG3 strain, at Day 672 | 0
  gp70-96ZM651.02 IgG3 strain, at Year 14 | 0
  gp70-BF1266_431a IgG3 strain, at Day 182 | 5
  gp70-BF1266_431a IgG3 strain, at Day 672 | 2
  gp70-BF1266_431a IgG3 strain, at Year 14 | 0
  gp70-BJOX002000.03.2 IgG3 strain, at Day 182 | 0
  gp70-BJOX002000.03.2 IgG3 strain, at Day 672 | 0
  gp70-BJOX002000.03.2 IgG3 strain, at Year 14 | 0
  gp70-C2101.c01 IgG3 strain, at Day 182 | 2
  gp70-C2101.c01 IgG3 strain, at Day 672 | 1
  gp70-C2101.c01 IgG3 strain, at Year 14 | 0
  gp70-CAP210.2.00.E8 IgG3 strain, at Day 182 | 0
  gp70-CAP210.2.00.E8 IgG3 strain, at Day 672 | 0
  gp70-CAP210.2.00.E8 IgG3 strain, at Year 14 | 0
  gp70-CM244.ec1 IgG3 strain, at Day 182 | 1
  gp70-CM244.ec1 IgG3 strain, at Day 672 | 0
  gp70-CM244.ec1 IgG3 strain, at Year 14 | 1
  gp70-Ce1086_B2 IgG3 strain, at Day 182 | 0
  gp70-Ce1086_B2 IgG3 strain, at Day 672 | 0
  gp70-Ce1086_B2 IgG3 strain, at Year 14 | 1
  gp70-RHPA4259.7 IgG3 strain, at Day 182 | 3
  gp70-RHPA4259.7 IgG3 strain, at Day 672 | 0
  gp70-RHPA4259.7 IgG3 strain, at Year 14 | 0
  gp70-TT31P.2F10.2792 IgG3 strain, at Day 182 | 2
  gp70-TT31P.2F10.2792 IgG3 strain, at Day 672 | 0
  gp70-TT31P.2F10.2792 IgG3 strain, at Year 14 | 0
  gp70-TV1.21 IgG3 strain, at Day 182: number analyzed (Participants) | 26
  gp70-TV1.21 IgG3 strain, at Day 182 | 3
  gp70-TV1.21 IgG3 strain, at Day 672: number analyzed (Participants) | 26
  gp70-TV1.21 IgG3 strain, at Day 672 | 0
  gp70-TV1.21 IgG3 strain, at Year 14: number analyzed (Participants) | 25
  gp70-TV1.21 IgG3 strain, at Year 14 | 0
  gp70_B.CaseA IgG3 strain, at Day 182: number analyzed (Participants) | 23
  gp70_B.CaseA IgG3 strain, at Day 182 | 11
  gp70_B.CaseA IgG3 strain, at Day 672: number analyzed (Participants) | 26
  gp70_B.CaseA IgG3 strain, at Day 672 | 2
  gp70_B.CaseA IgG3 strain, at Year 14: number analyzed (Participants) | 25
  gp70_B.CaseA IgG3 strain, at Year 14 | 0
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 182: number analyzed (Participants) | 28
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 182 | 15
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 672: number analyzed (Participants) | 28
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 672 | 5
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Year 14: number analyzed (Participants) | 27
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Year 14 | 2
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Day 182 | 1
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Day 672 | 1
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Year 14 | 1
  C.1086C_V1_V2 Tags IgG3 Qual strain, at Day 182 | 5
  C.1086C_V1_V2 Tags IgG3 Qual strain, at Day 672 | 0
  C.1086C_V1_V2 Tags IgG3 Qual strain, at Year 14 | 0
  C.1086C_V1_V2 Tags IgG4 Qual strain, at Day 182 | 0
  C.1086C_V1_V2 Tags IgG4 Qual strain, at Day 672 | 0
  C.1086C_V1_V2 Tags IgG4 Qual strain, at Year 14 | 0

4. Primary Outcome: Anti-V1V2 IgG1, IgG2, IgG3 and IgG4 Antibody BAMA Response Magnitude
Description: Whenever results were provided as "Mean Fluorescence Intensity (MFI)", the statistical outputs "BAMA response magnitude (MFI)" terminology is used instead of "concentrations/titres". Antigen IgG3 was assessed for all strains. Antigens IgG1, IgG2 and IgG4 were assessed only for C.1086C_V1_V2 Tags strain that was not part of any breadth panel. Due to low or infrequent response, or undetectable levels of response among the breadth panel strains, some additional strains, not part of the breadth panels, were also analyzed.
Time Frame: At Day 0, Day 182, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: MFI
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 34
MFI
  gp70-001428.2.42 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-001428.2.42 IgG3 strain, at Day 0 | 1.7 [1.1 to 2.6]
  gp70-001428.2.42 IgG3 strain, at Day 182 | 2.6 [1.5 to 4.4]
  gp70-001428.2.42 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-001428.2.42 IgG3 strain, at Day 672 | 1.5 [1.1 to 2.1]
  gp70-001428.2.42 IgG3 strain, at Year 14 | 1.4 [1.0 to 1.9]
  gp70-191084_B7 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-191084_B7 IgG3 strain, at Day 0 | 1.5 [1.1 to 2.1]
  gp70-191084_B7 IgG3 strain, at Day 182 | 4.6 [2.6 to 8.1]
  gp70-191084_B7 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-191084_B7 IgG3 strain, at Day 672 | 1.6 [1.1 to 2.6]
  gp70-191084_B7 IgG3 strain, at Year 14 | 2.8 [1.8 to 4.2]
  gp70-62357.14 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-62357.14 IgG3 strain, at Day 0 | 2.1 [1.4 to 3.2]
  gp70-62357.14 IgG3 strain, at Day 182 | 1.2 [1.0 to 1.4]
  gp70-62357.14 IgG3 strain, at Day 672 | 1.3 [1.0 to 1.6]
  gp70-62357.14 IgG3 strain, at Year 14 | 4.1 [2.8 to 6.0]
  gp70-700010058 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-700010058 IgG3 strain, at Day 0 | 1.2 [1.0 to 1.4]
  gp70-700010058 IgG3 strain, at Day 182 | 11.9 [6.3 to 22.6]
  gp70-700010058 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-700010058 IgG3 strain, at Day 672 | 1.3 [1.0 to 1.9]
  gp70-700010058 IgG3 strain, at Year 14 | 2.9 [1.9 to 4.2]
  gp70-7060101641 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-7060101641 IgG3 strain, at Day 0 | 1.1 [1.0 to 1.2]
  gp70-7060101641 IgG3 strain, at Day 182 | 3.7 [2.4 to 5.6]
  gp70-7060101641 IgG3 strain, at Day 672 | 1.4 [1.1 to 1.9]
  gp70-7060101641 IgG3 strain, at Year 14 | 1.0 [1.0 to 1.0]
  gp70-96ZM651.02 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-96ZM651.02 IgG3 strain, at Day 0 | 1.4 [1.0 to 2.0]
  gp70-96ZM651.02 IgG3 strain, at Day 182 | 1.8 [1.2 to 2.8]
  gp70-96ZM651.02 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-96ZM651.02 IgG3 strain, at Day 672 | 1.2 [0.9 to 1.6]
  gp70-96ZM651.02 IgG3 strain, at Year 14 | 1.6 [1.1 to 2.3]
  gp70-BF1266_431a IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-BF1266_431a IgG3 strain, at Day 0 | 1.0 [1.0 to 1.0]
  gp70-BF1266_431a IgG3 strain, at Day 182 | 13.2 [6.1 to 28.5]
  gp70-BF1266_431a IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-BF1266_431a IgG3 strain, at Day 672 | 1.8 [1.1 to 3.2]
  gp70-BF1266_431a IgG3 strain, at Year 14 | 1.5 [1.0 to 2.2]
  gp70-BJOX002000.03.2 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-BJOX002000.03.2 IgG3 strain, at Day 0 | 1.3 [1.0 to 1.6]
  gp70-BJOX002000.03.2 IgG3 strain, at Day 182 | 4.7 [2.9 to 7.7]
  gp70-BJOX002000.03.2 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-BJOX002000.03.2 IgG3 strain, at Day 672 | 1.3 [1.0 to 1.7]
  gp70-BJOX002000.03.2 IgG3 strain, at Year 14 | 1.6 [1.2 to 2.1]
  gp70-C2101.c01 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-C2101.c01 IgG3 strain, at Day 0 | 1.5 [0.9 to 2.5]
  gp70-C2101.c01 IgG3 strain, at Day 182 | 4.7 [2.4 to 9.1]
  gp70-C2101.c01 IgG3 strain, at Day 672 | 1.7 [1.0 to 3.0]
  gp70-C2101.c01 IgG3 strain, at Year 14 | 1.9 [1.2 to 3.0]
  gp70-CAP210.2.00.E8 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-CAP210.2.00.E8 IgG3 strain, at Day 0 | 1.5 [1.0 to 2.2]
  gp70-CAP210.2.00.E8 IgG3 strain, at Day 182 | 5.9 [3.6 to 9.5]
  gp70-CAP210.2.00.E8 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-CAP210.2.00.E8 IgG3 strain, at Day 672 | 1.6 [1.1 to 2.3]
  gp70-CAP210.2.00.E8 IgG3 strain, at Year 14 | 2.1 [1.5 to 3.1]
  gp70-CM244.ec1 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-CM244.ec1 IgG3 strain, at Day 0 | 1.5 [1.0 to 2.1]
  gp70-CM244.ec1 IgG3 strain, at Day 182 | 4.5 [2.7 to 7.6]
  gp70-CM244.ec1 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-CM244.ec1 IgG3 strain, at Day 672 | 1.5 [1.1 to 2.2]
  gp70-CM244.ec1 IgG3 strain, at Year 14 | 4.0 [2.5 to 6.5]
  gp70-Ce1086_B2 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-Ce1086_B2 IgG3 strain, at Day 0 | 1.7 [1.1 to 2.8]
  gp70-Ce1086_B2 IgG3 strain, at Day 182 | 3.0 [1.8 to 5.0]
  gp70-Ce1086_B2 IgG3 strain, at Day 672 | 1.4 [1.0 to 2.1]
  gp70-Ce1086_B2 IgG3 strain, at Year 14 | 1.4 [0.9 to 2.0]
  gp70-RHPA4259.7 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-RHPA4259.7 IgG3 strain, at Day 0 | 1.1 [0.9 to 1.3]
  gp70-RHPA4259.7 IgG3 strain, at Day 182 | 4.0 [2.0 to 7.9]
  gp70-RHPA4259.7 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-RHPA4259.7 IgG3 strain, at Day 672 | 1.0 [1.0 to 1.1]
  gp70-RHPA4259.7 IgG3 strain, at Year 14 | 1.2 [1.0 to 1.5]
  gp70-TT31P.2F10.2792 IgG3 strain, at Day 0: number analyzed (Participants) | 29
  gp70-TT31P.2F10.2792 IgG3 strain, at Day 0 | 1.3 [1.0 to 1.7]
  gp70-TT31P.2F10.2792 IgG3 strain, at Day 182 | 9.9 [5.7 to 16.9]
  gp70-TT31P.2F10.2792 IgG3 strain, at Day 672: number analyzed (Participants) | 33
  gp70-TT31P.2F10.2792 IgG3 strain, at Day 672 | 1.5 [1.1 to 2.1]
  gp70-TT31P.2F10.2792 IgG3 strain, at Year 14 | 1.1 [1.0 to 1.2]
  gp70-TV1.21 IgG3 strain, at Day 0: number analyzed (Participants) | 26
  gp70-TV1.21 IgG3 strain, at Day 0 | 1.6 [0.9 to 2.6]
  gp70-TV1.21 IgG3 strain, at Day 182: number analyzed (Participants) | 31
  gp70-TV1.21 IgG3 strain, at Day 182 | 11.4 [5.8 to 22.6]
  gp70-TV1.21 IgG3 strain, at Day 672: number analyzed (Participants) | 31
  gp70-TV1.21 IgG3 strain, at Day 672 | 1.9 [1.2 to 3.2]
  gp70-TV1.21 IgG3 strain, at Year 14: number analyzed (Participants) | 31
  gp70-TV1.21 IgG3 strain, at Year 14 | 2.9 [1.8 to 4.8]
  gp70_B.CaseA IgG3 strain, at Day 0: number analyzed (Participants) | 26
  gp70_B.CaseA IgG3 strain, at Day 0 | 1.2 [0.8 to 1.7]
  gp70_B.CaseA IgG3 strain, at Day 182: number analyzed (Participants) | 28
  gp70_B.CaseA IgG3 strain, at Day 182 | 58.2 [30.1 to 112.4]
  gp70_B.CaseA IgG3 strain, at Day 672: number analyzed (Participants) | 31
  gp70_B.CaseA IgG3 strain, at Day 672 | 2.8 [1.4 to 5.3]
  gp70_B.CaseA IgG3 strain, at Year 14: number analyzed (Participants) | 30
  gp70_B.CaseA IgG3 strain, at Year 14 | 1.7 [1.1 to 2.8]
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 0: number analyzed (Participants) | 28
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 0 | 1.2 [0.8 to 2.0]
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 182: number analyzed (Participants) | 33
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 182 | 89.4 [31.0 to 258.2]
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 672: number analyzed (Participants) | 33
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Day 672 | 7.4 [3.1 to 18.0]
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Year 14: number analyzed (Participants) | 32
  C.1086C_V1_V2 Tags IgG1 Qual strain, at Year 14 | 2.4 [1.3 to 4.7]
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Day 0: number analyzed (Participants) | 29
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Day 0 | 1.1 [1.0 to 1.2]
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Day 182: number analyzed (Participants) | 33
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Day 182 | 1.4 [0.9 to 2.1]
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Day 672: number analyzed (Participants) | 33
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Day 672 | 1.4 [0.9 to 2.1]
  C.1086C_V1_V2 Tags IgG2 Qual strain, at Year 14 | 1.3 [0.9 to 1.9]
  C.1086C_V1_V2 Tags IgG3 Qual strain, at Day 0: number analyzed (Participants) | 29
  C.1086C_V1_V2 Tags IgG3 Qual strain, at Day 0 | 1.8 [1.2 to 2.7]
  C.1086C_V1_V2 Tags IgG3 Qual strain, at Day 182 | 5.0 [2.2 to 11.1]
  C.1086C_V1_V2 Tags IgG3 Qual strain, at Day 672 | 1.3 [1.0 to 1.6]
  C.1086C_V1_V2 Tags IgG3 Qual strain, at Year 14 | 2.1 [1.6 to 2.8]
  C.1086C_V1_V2 Tags IgG4 Qual strain, at Day 0: number analyzed (Participants) | 29
  C.1086C_V1_V2 Tags IgG4 Qual strain, at Day 0 | 1.2 [1.0 to 1.4]
  C.1086C_V1_V2 Tags IgG4 Qual strain, at Day 182 | 1.3 [1.1 to 1.6]
  C.1086C_V1_V2 Tags IgG4 Qual strain, at Day 672 | 1.3 [1.1 to 1.6]
  C.1086C_V1_V2 Tags IgG4 Qual strain, at Year 14 | 1.0 [1.0 to 1.0]

5. Secondary Outcome: Number of Subjects With Anti-envelope Glycoprotein (Anti-gp) 120 Total IgG BAMA Response Call
Description: To comply with BAMA methodology and terminology, the wording "BAMA response call status" was used instead of "seropositivity" in the analysis. Compared to baseline result (Day 0), a sample is called "positive" for a given analyte if the response magnitude is equal to or above (≥) the analyte specific cutoff from all baseline samples in the study (where the cutoff is the 95th percentile of the baseline response, or 100, whichever is higher) OR ≥3 times the response magnitude as compared to the sample specific baseline. The strains: 086C_D7gp120.avi/293F IgG, Con 6 gp120/B IgG, and gp120 (Clone W6.1D) IgG were not part of any breadth panel. Due to low or infrequent response, or undetectable levels of response among the breadth panel strains, some additional strains, not part of the breadth panels, were also analyzed.
Time Frame: At Day 182, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 29
Participants
  254008_D11gp120.avi/293FIgGQual strain, at Day 182 | 29
  254008_D11gp120.avi/293FIgGQual strain, at Day 672 | 29
  254008_D11gp120.avi/293FIgGQual strain, at Year 14 | 27
  51802_D11gp120.avi/293F IgGQual strain, at Day 182: number analyzed (Participants) | 27
  51802_D11gp120.avi/293F IgGQual strain, at Day 182 | 25
  51802_D11gp120.avi/293F IgGQual strain, at Day 672: number analyzed (Participants) | 27
  51802_D11gp120.avi/293F IgGQual strain, at Day 672 | 18
  51802_D11gp120.avi/293F IgGQual strain, at Year 14: number analyzed (Participants) | 22
  51802_D11gp120.avi/293F IgGQual strain, at Year 14 | 6
  A244 D11gp120_avi IgG Qual strain, at Day 182: number analyzed (Participants) | 27
  A244 D11gp120_avi IgG Qual strain, at Day 182 | 25
  A244 D11gp120_avi IgG Qual strain, at Day 672: number analyzed (Participants) | 27
  A244 D11gp120_avi IgG Qual strain, at Day 672 | 20
  A244 D11gp120_avi IgG Qual strain, at Year 14: number analyzed (Participants) | 22
  A244 D11gp120_avi IgG Qual strain, at Year 14 | 8
  B.6240_D11gp120/293F IgG Qual strain, at Day 182: number analyzed (Participants) | 27
  B.6240_D11gp120/293F IgG Qual strain, at Day 182 | 27
  B.6240_D11gp120/293F IgG Qual strain, at Day 672: number analyzed (Participants) | 27
  B.6240_D11gp120/293F IgG Qual strain, at Day 672 | 23
  B.6240_D11gp120/293F IgG Qual strain, at Year 14: number analyzed (Participants) | 22
  B.6240_D11gp120/293F IgG Qual strain, at Year 14 | 17
  BJOX002_D11gp120.avi/293FIgGQual strain,at Day 182: number analyzed (Participants) | 27
  BJOX002_D11gp120.avi/293FIgGQual strain,at Day 182 | 21
  BJOX002_D11gp120.avi/293FIgGQual strain,at Day 672: number analyzed (Participants) | 27
  BJOX002_D11gp120.avi/293FIgGQual strain,at Day 672 | 13
  BJOX002_D11gp120.avi/293FIgGQual strain,at Year 14: number analyzed (Participants) | 22
  BJOX002_D11gp120.avi/293FIgGQual strain,at Year 14 | 2
  BORI_D11gp120.avi/293F IgG Qual strain, at Day 182: number analyzed (Participants) | 27
  BORI_D11gp120.avi/293F IgG Qual strain, at Day 182 | 26
  BORI_D11gp120.avi/293F IgG Qual strain, at Day 672: number analyzed (Participants) | 27
  BORI_D11gp120.avi/293F IgG Qual strain, at Day 672 | 20
  BORI_D11gp120.avi/293F IgG Qual strain, at Year 14: number analyzed (Participants) | 22
  BORI_D11gp120.avi/293F IgG Qual strain, at Year 14 | 10
  CNE20_D11gp120.avi/293F IgGQual strain, at Day 182: number analyzed (Participants) | 27
  CNE20_D11gp120.avi/293F IgGQual strain, at Day 182 | 26
  CNE20_D11gp120.avi/293F IgGQual strain, at Day 672: number analyzed (Participants) | 27
  CNE20_D11gp120.avi/293F IgGQual strain, at Day 672 | 23
  CNE20_D11gp120.avi/293F IgGQual strain, at Year 14: number analyzed (Participants) | 22
  CNE20_D11gp120.avi/293F IgGQual strain, at Year 14 | 16
  TT31P.2792_D11gp120.avi/293FIgGQual, at Day 182: number analyzed (Participants) | 27
  TT31P.2792_D11gp120.avi/293FIgGQual, at Day 182 | 27
  TT31P.2792_D11gp120.avi/293FIgGQual, at Day 672: number analyzed (Participants) | 27
  TT31P.2792_D11gp120.avi/293FIgGQual, at Day 672 | 26
  TT31P.2792_D11gp120.avi/293FIgGQual, at Year 14: number analyzed (Participants) | 22
  TT31P.2792_D11gp120.avi/293FIgGQual, at Year 14 | 20
  1086C_D7gp120.avi/293F IgG strain, at Day 182: number analyzed (Participants) | 27
  1086C_D7gp120.avi/293F IgG strain, at Day 182 | 27
  1086C_D7gp120.avi/293F IgG strain, at Day 672: number analyzed (Participants) | 27
  1086C_D7gp120.avi/293F IgG strain, at Day 672 | 27
  1086C_D7gp120.avi/293F IgG strain, at Year 14: number analyzed (Participants) | 22
  1086C_D7gp120.avi/293F IgG strain, at Year 14 | 22
  Con 6 gp120/B IgG strain, at Day 182: number analyzed (Participants) | 27
  Con 6 gp120/B IgG strain, at Day 182 | 27
  Con 6 gp120/B IgG strain, at Day 672: number analyzed (Participants) | 27
  Con 6 gp120/B IgG strain, at Day 672 | 25
  Con 6 gp120/B IgG strain, at Year 14: number analyzed (Participants) | 22
  Con 6 gp120/B IgG strain, at Year 14 | 16
  gp120 (Clone W6.1D) IgG strain, at Day 182: number analyzed (Participants) | 27
  gp120 (Clone W6.1D) IgG strain, at Day 182 | 27
  gp120 (Clone W6.1D) IgG strain, at Day 672: number analyzed (Participants) | 27
  gp120 (Clone W6.1D) IgG strain, at Day 672 | 25
  gp120 (Clone W6.1D) IgG strain, at Year 14: number analyzed (Participants) | 22
  gp120 (Clone W6.1D) IgG strain, at Year 14 | 19

6. Secondary Outcome: Anti-gp 120 Total IgG Antibody BAMA Response Magnitude
Description: Whenever results were provided as "Mean Fluorescence Intensity (MFI)", the statistical outputs "BAMA response magnitude (MFI)" terminology is used instead of "concentrations/titres". The strains: 086C_D7gp120.avi/293F IgG, Con 6 gp120/B IgG, and gp120 (Clone W6.1D) IgG were not part of any breadth panel. Due to low or infrequent response, or undetectable levels of response among the breadth panel strains, some additional strains, not part of the breadth panels, were also analyzed.
Time Frame: At Day 0, Day 182, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: MFI
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 34
MFI
  254008_D11gp120.avi/293F IgG -BKG strain, at Day 0: number analyzed (Participants) | 29
  254008_D11gp120.avi/293F IgG -BKG strain, at Day 0 | 2.5 [1.4 to 4.4]
  254008_D11gp120.avi/293FIgGQual strain, at Day 182 | 6796.7 [5926.0 to 7795.3]
  254008_D11gp120.avi/293FIgGQual strain, at day 672 | 1633.3 [1361.1 to 1959.9]
  254008_D11gp120.avi/293FIgGQual strain, at Year 14 | 479.6 [308.7 to 745.3]
  51802_D11gp120.avi/293F IgG -BKG strain, at Day 0: number analyzed (Participants) | 27
  51802_D11gp120.avi/293F IgG -BKG strain, at Day 0 | 1.0 [1.0 to 1.0]
  51802_D11gp120.avi/293F IgGQual strain, at Day 182: number analyzed (Participants) | 32
  51802_D11gp120.avi/293F IgGQual strain, at Day 182 | 993.7 [407.4 to 2424.1]
  51802_D11gp120.avi/293F IgGQual strain, at Day 672: number analyzed (Participants) | 31
  51802_D11gp120.avi/293F IgGQual strain, at Day 672 | 74.8 [29.0 to 193.3]
  51802_D11gp120.avi/293F IgGQual strain, at Year 14: number analyzed (Participants) | 26
  51802_D11gp120.avi/293F IgGQual strain, at Year 14 | 14.4 [5.7 to 36.4]
  A244 D11gp120_avi IgG -BKG strain, at Day 0: number analyzed (Participants) | 27
  A244 D11gp120_avi IgG -BKG strain, at Day 0 | 1.4 [0.9 to 2.2]
  A244 D11gp120_avi IgG Qual strain, at Day 182: number analyzed (Participants) | 32
  A244 D11gp120_avi IgG Qual strain, at Day 182 | 990.2 [498.3 to 1967.7]
  A244 D11gp120_avi IgG Qual strain, at Day 672: number analyzed (Participants) | 31
  A244 D11gp120_avi IgG Qual strain, at Day 672 | 124.4 [50.2 to 308.2]
  A244 D11gp120_avi IgG Qual strain, at Year 14: number analyzed (Participants) | 26
  A244 D11gp120_avi IgG Qual strain, at Year 14 | 39.8 [17.6 to 90.2]
  B.6240_D11gp120/293F IgG -BKG strain, at Day 0: number analyzed (Participants) | 27
  B.6240_D11gp120/293F IgG -BKG strain, at Day 0 | 1.0 [1.0 to 1.0]
  B.6240_D11gp120/293F IgG Qual strain, at Day 182: number analyzed (Participants) | 32
  B.6240_D11gp120/293F IgG Qual strain, at Day 182 | 8760.5 [6725.8 to 11410.7]
  B.6240_D11gp120/293F IgG Qual strain, at Day 672: number analyzed (Participants) | 31
  B.6240_D11gp120/293F IgG Qual strain, at Day 672 | 634.2 [265.8 to 1513.3]
  B.6240_D11gp120/293F IgG Qual strain, at Year 14: number analyzed (Participants) | 26
  B.6240_D11gp120/293F IgG Qual strain, at Year 14 | 132.8 [53.6 to 329.1]
  BJOX002_D11gp120.avi/293F IgG-BKG strain, at Day 0: number analyzed (Participants) | 27
  BJOX002_D11gp120.avi/293F IgG-BKG strain, at Day 0 | 1.1 [0.9 to 1.3]
  BJOX002_D11gp120.avi/293FIgGQual strain,at Day 182: number analyzed (Participants) | 32
  BJOX002_D11gp120.avi/293FIgGQual strain,at Day 182 | 250.6 [109.9 to 571.6]
  BJOX002_D11gp120.avi/293FIgGQual strain,at Day 672: number analyzed (Participants) | 31
  BJOX002_D11gp120.avi/293FIgGQual strain,at Day 672 | 31.2 [13.8 to 70.6]
  BJOX002_D11gp120.avi/293FIgGQual strain,at Year 14: number analyzed (Participants) | 26
  BJOX002_D11gp120.avi/293FIgGQual strain,at Year 14 | 9.9 [4.5 to 21.9]
  BORI_D11gp120.avi/293F IgG -BKG strain, at Day 0: number analyzed (Participants) | 27
  BORI_D11gp120.avi/293F IgG -BKG strain, at Day 0 | 1.0 [1.0 to 1.0]
  BORI_D11gp120.avi/293F IgG Qual strain, at Day 182: number analyzed (Participants) | 32
  BORI_D11gp120.avi/293F IgG Qual strain, at Day 182 | 2811.9 [1546.5 to 5112.6]
  BORI_D11gp120.avi/293F IgG Qual strain, at Day 672: number analyzed (Participants) | 31
  BORI_D11gp120.avi/293F IgG Qual strain, at Day 672 | 148.9 [57.1 to 388.5]
  BORI_D11gp120.avi/293F IgG Qual strain, at Year 14: number analyzed (Participants) | 26
  BORI_D11gp120.avi/293F IgG Qual strain, at Year 14 | 35.5 [13.8 to 91.4]
  CNE20_D11gp120.avi/293F IgG -BKG strain, at Day 0: number analyzed (Participants) | 27
  CNE20_D11gp120.avi/293F IgG -BKG strain, at Day 0 | 1.1 [0.9 to 1.5]
  CNE20_D11gp120.avi/293F IgGQual strain, at Day 182: number analyzed (Participants) | 32
  CNE20_D11gp120.avi/293F IgGQual strain, at Day 182 | 2925.8 [1336.2 to 6406.5]
  CNE20_D11gp120.avi/293F IgGQual strain, at Day 672: number analyzed (Participants) | 31
  CNE20_D11gp120.avi/293F IgGQual strain, at Day 672 | 587.3 [295.6 to 1166.9]
  CNE20_D11gp120.avi/293F IgGQual strain, at Year 14: number analyzed (Participants) | 26
  CNE20_D11gp120.avi/293F IgGQual strain, at Year 14 | 126.0 [55.6 to 285.5]
  TT31P.2792_D11gp120.avi/293FIgGBKG strain,at Day 0: number analyzed (Participants) | 27
  TT31P.2792_D11gp120.avi/293FIgGBKG strain,at Day 0 | 1.6 [0.9 to 2.7]
  TT31P.2792_D11gp120.avi/293FIgGQual, at Day 182: number analyzed (Participants) | 32
  TT31P.2792_D11gp120.avi/293FIgGQual, at Day 182 | 20622.9 [18541.3 to 22938.2]
  TT31P.2792_D11gp120.avi/293FIgGQual, at Day 672: number analyzed (Participants) | 31
  TT31P.2792_D11gp120.avi/293FIgGQual, at Day 672 | 3372.5 [1788.3 to 6360.1]
  TT31P.2792_D11gp120.avi/293FIgGQual, at Year 14: number analyzed (Participants) | 26
  TT31P.2792_D11gp120.avi/293FIgGQual, at Year 14 | 568.6 [253.3 to 1276.5]
  1086C_D7gp120.avi/293F IgG strain, at Day 0: number analyzed (Participants) | 27
  1086C_D7gp120.avi/293F IgG strain, at Day 0 | 1.1 [0.9 to 1.4]
  1086C_D7gp120.avi/293F IgG strain, at Day 182: number analyzed (Participants) | 32
  1086C_D7gp120.avi/293F IgG strain, at Day 182 | 27145.5 [26416.5 to 27894.7]
  1086C_D7gp120.avi/293F IgG strain, at Day 672: number analyzed (Participants) | 31
  1086C_D7gp120.avi/293F IgG strain, at Day 672 | 17448.6 [14249.1 to 21366.6]
  1086C_D7gp120.avi/293F IgG strain, at Year 14: number analyzed (Participants) | 26
  1086C_D7gp120.avi/293F IgG strain, at Year 14 | 4253.8 [3218.3 to 5622.4]
  Con 6 gp120/B IgG strain, at Day 0: number analyzed (Participants) | 27
  Con 6 gp120/B IgG strain, at Day 0 | 1.8 [1.2 to 2.6]
  Con 6 gp120/B IgG strain, at Day 182: number analyzed (Participants) | 32
  Con 6 gp120/B IgG strain, at Day 182 | 10618.0 [8540.0 to 13201.6]
  Con 6 gp120/B IgG strain, at Day 672: number analyzed (Participants) | 31
  Con 6 gp120/B IgG strain, at Day 672 | 879.2 [422.1 to 1831.4]
  Con 6 gp120/B IgG strain, at Year 14: number analyzed (Participants) | 26
  Con 6 gp120/B IgG strain, at Year 14 | 176.8 [76.6 to 408.1]
  gp120 (Clone W6.1D) IgG strain, at Day 0: number analyzed (Participants) | 27
  gp120 (Clone W6.1D) IgG strain, at Day 0 | 1.1 [0.9 to 1.3]
  gp120 (Clone W6.1D) IgG strain, at Day 182: number analyzed (Participants) | 32
  gp120 (Clone W6.1D) IgG strain, at Day 182 | 25617.4 [24497.6 to 26788.4]
  gp120 (Clone W6.1D) IgG strain, at Day 672: number analyzed (Participants) | 31
  gp120 (Clone W6.1D) IgG strain, at Day 672 | 3027.1 [1293.7 to 7083.2]
  gp120 (Clone W6.1D) IgG strain, at Year 14: number analyzed (Participants) | 26
  gp120 (Clone W6.1D) IgG strain, at Year 14 | 544.6 [236.5 to 1253.7]

7. Secondary Outcome: Number of Subjects With Anti-gp120 (IgG1, IgG2, IgG3 and IgG4) BAMA Response Call for Analytes Not Part of Any Breadth Panel
Description: To comply with BAMA methodology and terminology, the wording "BAMA response call status" was used instead of "seropositivity" in the analysis. Compared to baseline result (Day 0), a sample is called "positive" for a given analyte if the response magnitude is equal to or above (≥) the analyte specific cutoff from all baseline samples in the study (where the cutoff is the 95th percentile of the baseline response, or 100, whichever is higher) OR ≥3 times the response magnitude as compared to the sample specific baseline.Analysis was performed on the gp120 antigen (IgG1, IgG2, IgG3 and IgG4) for the following vaccine HIV strains which were not part of any breadth panel: 1086C_D7gp120.avi/293F IgG, Con 6 gp120/B IgG, and gp120 (Clone W6.1D) IgG. Due to low or infrequent response, or undetectable levels of response among the breadth panel strains, some additional strains, not part of the breadth panels, were also analyzed.
Time Frame: At Day 182, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 29
Participants
  1086C_D7gp120.avi/293F IgG1 strain, at Day 182: number analyzed (Participants) | 28
  1086C_D7gp120.avi/293F IgG1 strain, at Day 182 | 28
  1086C_D7gp120.avi/293F IgG1 strain, at Day 672: number analyzed (Participants) | 28
  1086C_D7gp120.avi/293F IgG1 strain, at Day 672 | 27
  1086C_D7gp120.avi/293F IgG1 strain, at Year 14: number analyzed (Participants) | 27
  1086C_D7gp120.avi/293F IgG1 strain, at Year 14 | 23
  Con 6 gp120/B IgG1 strain, at Day 182: number analyzed (Participants) | 28
  Con 6 gp120/B IgG1 strain, at Day 182 | 28
  Con 6 gp120/B IgG1 strain, at Day 672: number analyzed (Participants) | 28
  Con 6 gp120/B IgG1 strain, at Day 672 | 22
  Con 6 gp120/B IgG1 strain, at Year 14: number analyzed (Participants) | 27
  Con 6 gp120/B IgG1 strain, at Year 14 | 11
  gp120 (Clone W6.1D) IgG1 strain, at Day 182: number analyzed (Participants) | 28
  gp120 (Clone W6.1D) IgG1 strain, at Day 182 | 28
  gp120 (Clone W6.1D) IgG1 strain, at Day 672: number analyzed (Participants) | 28
  gp120 (Clone W6.1D) IgG1 strain, at Day 672 | 25
  gp120 (Clone W6.1D) IgG1 strain, at Year 14: number analyzed (Participants) | 27
  gp120 (Clone W6.1D) IgG1 strain, at Year 14 | 16
  1086C_D7gp120.avi/293F IgG2 strain, at Day 182 | 0
  1086C_D7gp120.avi/293F IgG2 strain, at Day 672 | 0
  1086C_D7gp120.avi/293F IgG2 strain, at Year 14 | 0
  Con 6 gp120/B IgG2 strain, at Day 182 | 0
  Con 6 gp120/B IgG2 strain, at Day 672 | 0
  Con 6 gp120/B IgG2 strain, at Year 14 | 0
  gp120 (Clone W6.1D) IgG2 strain, at Day 182 | 0
  gp120 (Clone W6.1D) IgG2 strain, at Day 672 | 0
  gp120 (Clone W6.1D) IgG2 strain, at Year 14 | 0
  1086C_D7gp120.avi/293F IgG3 strain, at Day 182: number analyzed (Participants) | 26
  1086C_D7gp120.avi/293F IgG3 strain, at Day 182 | 25
  1086C_D7gp120.avi/293F IgG3 strain, at Day 672: number analyzed (Participants) | 26
  1086C_D7gp120.avi/293F IgG3 strain, at Day 672 | 21
  1086C_D7gp120.avi/293F IgG3 strain, at Year 14: number analyzed (Participants) | 25
  1086C_D7gp120.avi/293F IgG3 strain, at Year 14 | 9
  Con 6 gp120/B IgG3 strain, at Day 182: number analyzed (Participants) | 26
  Con 6 gp120/B IgG3 strain, at Day 182 | 9
  Con 6 gp120/B IgG3 strain, at Day 672: number analyzed (Participants) | 26
  Con 6 gp120/B IgG3 strain, at Day 672 | 0
  Con 6 gp120/B IgG3 strain, at Year 14: number analyzed (Participants) | 25
  Con 6 gp120/B IgG3 strain, at Year 14 | 0
  gp120 (Clone W6.1D) IgG3 strain, at Day 182: number analyzed (Participants) | 26
  gp120 (Clone W6.1D) IgG3 strain, at Day 182 | 19
  gp120 (Clone W6.1D) IgG3 strain, at Day 672: number analyzed (Participants) | 26
  gp120 (Clone W6.1D) IgG3 strain, at Day 672 | 3
  gp120 (Clone W6.1D) IgG3 strain, at Year 14: number analyzed (Participants) | 25
  gp120 (Clone W6.1D) IgG3 strain, at Year 14 | 1
  1086C_D7gp120.avi/293F IgG4 strain, at Day 182 | 6
  1086C_D7gp120.avi/293F IgG4 strain, at Day 672 | 5
  1086C_D7gp120.avi/293F IgG4 strain, at Year 14 | 7
  Con 6 gp120/B IgG4 strain, at Day 182 | 1
  Con 6 gp120/B IgG4 strain, at Day 672 | 2
  Con 6 gp120/B IgG4 strain, at Year 14 | 2
  gp120 (Clone W6.1D) IgG4 strain, at Day 182 | 8
  gp120 (Clone W6.1D) IgG4 strain, at Day 672 | 3
  gp120 (Clone W6.1D) IgG4 strain, at Year 14 | 3

8. Secondary Outcome: Anti-gp120 (IgG1, IgG2, IgG3 and IgG4) BAMA Response Magnitude for Analytes Not Part of Any Breadth Panel
Description: Whenever results were provided as "Mean Fluorescence Intensity (MFI)", the statistical outputs "BAMA response magnitude (MFI)" terminology is used instead of "concentrations/titres". Analysis was performed on the gp120 antigen (IgG1, IgG2, IgG3 and IgG4) for the following vaccine HIV strains: which were not part of any breadth panel: 1086C_D7gp120.avi/293F IgG, Con 6 gp120/B IgG, and gp120 (Clone W6.1D) IgG. Due to low or infrequent response, or undetectable levels of response among the breadth panel strains, some additional strains, not part of the breadth panels, were also analyzed.
Time Frame: At Day 0, Day 182, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: MFI
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 34
MFI
  1086C_D7gp120.avi/293F IgG1 strain, at Day 0: number analyzed (Participants) | 28
  1086C_D7gp120.avi/293F IgG1 strain, at Day 0 | 1.0 [1.0 to 1.0]
  1086C_D7gp120.avi/293F IgG1 strain, at Day 182: number analyzed (Participants) | 33
  1086C_D7gp120.avi/293F IgG1 strain, at Day 182 | 10365.4 [9153.8 to 11737.5]
  1086C_D7gp120.avi/293F IgG1 strain, at Day 672: number analyzed (Participants) | 33
  1086C_D7gp120.avi/293F IgG1 strain, at Day 672 | 2834.1 [1991.6 to 4033.1]
  1086C_D7gp120.avi/293F IgG1 strain, at Year 14: number analyzed (Participants) | 32
  1086C_D7gp120.avi/293F IgG1 strain, at Year 14 | 371.0 [158.9 to 866.0]
  Con 6 gp120/B IgG1 strain, at Day 0: number analyzed (Participants) | 28
  Con 6 gp120/B IgG1 strain, at Day 0 | 1.0 [1.0 to 1.1]
  Con 6 gp120/B IgG1 strain, at Day 182: number analyzed (Participants) | 33
  Con 6 gp120/B IgG1 strain, at Day 182 | 4396.8 [3618.2 to 5343.0]
  Con 6 gp120/B IgG1 strain, at Day 672: number analyzed (Participants) | 33
  Con 6 gp120/B IgG1 strain, at Day 672 | 246.0 [95.6 to 632.9]
  Con 6 gp120/B IgG1 strain, at Year 14: number analyzed (Participants) | 32
  Con 6 gp120/B IgG1 strain, at Year 14 | 21.5 [8.2 to 55.9]
  gp120 (Clone W6.1D) IgG1 strain, at Day 0: number analyzed (Participants) | 28
  gp120 (Clone W6.1D) IgG1 strain, at Day 0 | 1.0 [1.0 to 1.0]
  gp120 (Clone W6.1D) IgG1 strain, at Day 182: number analyzed (Participants) | 33
  gp120 (Clone W6.1D) IgG1 strain, at Day 182 | 11572.9 [9525.5 to 14060.3]
  gp120 (Clone W6.1D) IgG1 strain, at Day 672: number analyzed (Participants) | 33
  gp120 (Clone W6.1D) IgG1 strain, at Day 672 | 653.3 [359.5 to 1187.2]
  gp120 (Clone W6.1D) IgG1 strain, at Year 14: number analyzed (Participants) | 32
  gp120 (Clone W6.1D) IgG1 strain, at Year 14 | 47.0 [18.1 to 122.1]
  1086C_D7gp120.avi/293F IgG2 strain, at Day 0: number analyzed (Participants) | 29
  1086C_D7gp120.avi/293F IgG2 strain, at Day 0 | 1.2 [1.1 to 1.4]
  1086C_D7gp120.avi/293F IgG2 strain, at Day 182: number analyzed (Participants) | 33
  1086C_D7gp120.avi/293F IgG2 strain, at Day 182 | 2.6 [1.7 to 3.9]
  1086C_D7gp120.avi/293F IgG2 strain, at Day 672: number analyzed (Participants) | 33
  1086C_D7gp120.avi/293F IgG2 strain, at Day 672 | 2.4 [1.6 to 3.6]
  1086C_D7gp120.avi/293F IgG2 strain, at Year 14 | 1.1 [1.0 to 1.2]
  Con 6 gp120/B IgG2 strain, at Day 0: number analyzed (Participants) | 29
  Con 6 gp120/B IgG2 strain, at Day 0 | 1.1 [1.0 to 1.2]
  Con 6 gp120/B IgG2 strain, at Day 182: number analyzed (Participants) | 33
  Con 6 gp120/B IgG2 strain, at Day 182 | 1.3 [1.1 to 1.6]
  Con 6 gp120/B IgG2 strain, at Day 672: number analyzed (Participants) | 33
  Con 6 gp120/B IgG2 strain, at Day 672 | 1.4 [1.1 to 1.7]
  Con 6 gp120/B IgG2 strain, at Year 14 | 1.3 [1.1 to 1.6]
  gp120 (Clone W6.1D) IgG2 strain, at Day 0: number analyzed (Participants) | 29
  gp120 (Clone W6.1D) IgG2 strain, at Day 0 | 1.0 [1.0 to 1.0]
  gp120 (Clone W6.1D) IgG2 strain, at Day 182: number analyzed (Participants) | 33
  gp120 (Clone W6.1D) IgG2 strain, at Day 182 | 1.9 [1.3 to 2.9]
  gp120 (Clone W6.1D) IgG2 strain, at Day 672: number analyzed (Participants) | 33
  gp120 (Clone W6.1D) IgG2 strain, at Day 672 | 1.5 [1.1 to 2.0]
  gp120 (Clone W6.1D) IgG2 strain, at Year 14 | 1.1 [0.9 to 1.4]
  1086C_D7gp120.avi/293F IgG3 strain, at Day 0: number analyzed (Participants) | 26
  1086C_D7gp120.avi/293F IgG3 strain, at Day 0 | 1.5 [1.1 to 2.0]
  1086C_D7gp120.avi/293F IgG3 strain, at Day 182: number analyzed (Participants) | 31
  1086C_D7gp120.avi/293F IgG3 strain, at Day 182 | 417.1 [302.7 to 574.8]
  1086C_D7gp120.avi/293F IgG3 strain, at Day 672: number analyzed (Participants) | 31
  1086C_D7gp120.avi/293F IgG3 strain, at Day 672 | 206.3 [150.4 to 283.1]
  1086C_D7gp120.avi/293F IgG3 strain, at Year 14: number analyzed (Participants) | 30
  1086C_D7gp120.avi/293F IgG3 strain, at Year 14 | 42.8 [22.4 to 81.8]
  Con 6 gp120/B IgG3 strain, at Day 0: number analyzed (Participants) | 26
  Con 6 gp120/B IgG3 strain, at Day 0 | 1.1 [1.0 to 1.2]
  Con 6 gp120/B IgG3 strain, at Day 182: number analyzed (Participants) | 31
  Con 6 gp120/B IgG3 strain, at Day 182 | 60.8 [41.5 to 89.0]
  Con 6 gp120/B IgG3 strain, at Day 672: number analyzed (Participants) | 31
  Con 6 gp120/B IgG3 strain, at Day 672 | 11.0 [6.5 to 18.6]
  Con 6 gp120/B IgG3 strain, at Year 14: number analyzed (Participants) | 30
  Con 6 gp120/B IgG3 strain, at Year 14 | 2.9 [1.9 to 4.3]
  gp120 (Clone W6.1D) IgG3 strain, at Day 0: number analyzed (Participants) | 26
  gp120 (Clone W6.1D) IgG3 strain, at Day 0 | 1.1 [1.0 to 1.2]
  gp120 (Clone W6.1D) IgG3 strain, at Day 182: number analyzed (Participants) | 31
  gp120 (Clone W6.1D) IgG3 strain, at Day 182 | 161.9 [111.2 to 235.6]
  gp120 (Clone W6.1D) IgG3 strain, at Day 672: number analyzed (Participants) | 31
  gp120 (Clone W6.1D) IgG3 strain, at Day 672 | 24.3 [14.7 to 40.3]
  gp120 (Clone W6.1D) IgG3 strain, at Year 14: number analyzed (Participants) | 30
  gp120 (Clone W6.1D) IgG3 strain, at Year 14 | 7.8 [4.3 to 14.3]
  1086C_D7gp120.avi/293F IgG4 strain, at Day 0: number analyzed (Participants) | 29
  1086C_D7gp120.avi/293F IgG4 strain, at Day 0 | 1.2 [1.0 to 1.4]
  1086C_D7gp120.avi/293F IgG4 strain, at Day 182 | 47.0 [30.4 to 72.7]
  1086C_D7gp120.avi/293F IgG4 strain, at Day 672 | 30.1 [16.9 to 53.6]
  1086C_D7gp120.avi/293F IgG4 strain, at Year 14 | 20.3 [9.9 to 41.5]
  Con 6 gp120/B IgG4 strain, at Day 0: number analyzed (Participants) | 29
  Con 6 gp120/B IgG4 strain, at Day 0 | 1.0 [1.0 to 1.0]
  Con 6 gp120/B IgG4 strain, at Day 182 | 14.9 [9.7 to 22.7]
  Con 6 gp120/B IgG4 strain, at Day 672 | 6.6 [3.9 to 11.3]
  Con 6 gp120/B IgG4 strain, at Year 14 | 4.7 [2.5 to 8.6]
  gp120 (Clone W6.1D) IgG4 strain, at Day 0: number analyzed (Participants) | 29
  gp120 (Clone W6.1D) IgG4 strain, at Day 0 | 1.1 [1.0 to 1.2]
  gp120 (Clone W6.1D) IgG4 strain, at Day 182 | 52.8 [36.7 to 75.8]
  gp120 (Clone W6.1D) IgG4 strain, at Day 672 | 21.3 [12.9 to 35.3]
  gp120 (Clone W6.1D) IgG4 strain, at Year 14 | 10.4 [5.8 to 18.8]

9. Secondary Outcome: Frequency of Human Immunodeficiency Virus Type 1 (HIV-1) Specific Cluster of Differentiation-4 (CD4+) T Cells Expressing at Least 2 Cytokine Markers
Description: Assessed cytokines include: cluster of differentiation-40 lingand (CD40-L), Interleukin-2 (IL2), Tumour Necrosis Factor-alpha (TNF-α), Interferon-gamma (INF-γ), by Intracellular Cytokine Staining (ICS). CD4+ T-cells were expressed in CD4+ T-cells/million cells.
Time Frame: At Day 0, Day 98, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 33
CD4+ T-cells/million cells
  At Day 0: number analyzed (Participants) | 26
  At Day 0 | 0.00 [0.00 to 0.01]
  At Day 98 | 0.42 [0.30 to 0.78]
  At Day 672: number analyzed (Participants) | 30
  At Day 672 | 0.32 [0.21 to 0.43]
  At Year 14: number analyzed (Participants) | 32
  At Year 14 | 0.21 [0.14 to 0.35]

10. Secondary Outcome: Number of Vaccine Responders for HIV-1-specific CD4+ T-cells Expressing at Least 2 Cytokine Markers
Description: Vaccine response rates for HIV-1-specific CD4+ T cells expressing at least two markers among CD40L, IL-2, TNF-α and IFN-γ with responders were defined as subjects with: a 2-fold increase as compared to the cut-off (=354, limit of quantification [LOQ] of the assay), for subjects with pre-vaccination frequency below the cut-off, at Day 0, OR at least 2-fold increase as compared to pre-vaccination frequency, for subjects with pre-vaccination frequency above the cut-off.
Time Frame: At Day 98 and at Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 26
Participants
  At Day 98 | 25
  At Day 672: number analyzed (Participants) | 23
  At Day 672 | 23
  At Year 14: number analyzed (Participants) | 24
  At Year 14 | 22

11. Secondary Outcome: Frequency of Human Immunodeficiency Virus Type 1 (HIV-1) Specific CD8+ T-cells Expressing at Least 2 Cytokine Markers
Description: Assessed cytokines include: CD40-L, IL2, TNF-α, INF-γ, by ICS. CD8+ T-cells were expressed in CD8+ T-cells/million cells/million cells.
Time Frame: At Day 0, Day 98, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 33
CD8+ T-cells/million cells
  At Day 0: number analyzed (Participants) | 27
  At Day 0 | 0.00 [0.00 to 0.01]
  At Day 98: number analyzed (Participants) | 31
  At Day 98 | 0.00 [0.00 to 0.01]
  At Day 672: number analyzed (Participants) | 32
  At Day 672 | 0.00 [0.00 to 0.01]
  At Year 14 | 0.00 [0.00 to 0.01]

12. Secondary Outcome: Number of Vaccine Responders for HIV-1-specific CD8+ T-cells Expressing at Least 2 Cytokine Markers
Description: Vaccine response rates for HIV-1-specific CD8+ T cells expressing at least two markers among CD40L, IL-2, TNF-α and IFN-γ with responders were defined as subjects with: a 2-fold increase as compared to the cut-off (=354, limit of quantification [LOQ] of the assay), for subjects with pre-vaccination frequency below the cut-off, at Day 0, OR at least 2-fold increase as compared to pre- vaccination frequency, for subjects with pre-vaccination frequency above the cut-off.
Time Frame: At Day 98, Day 672 historical time points of PRO-HIV-002 and at Year 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSKSB732461 Group
Number analyzed (Participants) | 33
Participants
  At Day 98 | 0
  At Day 672 | 0
  At Year 14 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were reported during the whole study period (single study visit, at Year 14). Adverse events were not collected.
Description: Only SAEs related to study participation or to a concurrent GSK medication/product were collected and recorded from the time the subject consented to participate in the study (i.e., ICF signature) until the subject was discharged from the study.
Arm/Group | GSKSB732461 Group
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03368053/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT03368053/SAP_001.pdf